CLINICAL TRIAL: NCT05968313
Title: Abnormal Neural Pain Empathic Processing in Adolescents With Non-suicidal Self-Injury
Brief Title: Altered Neural Pain Empathic Reactivity in NSSI Adolescents
Status: Recruiting | Type: Observational
Sponsor: University of Electronic Science and Technology of China (Other)
Responsible Party: Principal Investigator, Benjamin Becker, Professor, University of Electronic Science and Technology of China
Other Study IDs: BAM_lab_NSSI_02
Record Dates: First submitted 2023-07-20; First posted 2023-08-01 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Nonsuicidal Self Injury; Pain Empathy
MeSH Terms: conditions — Self-Injurious Behavior

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- NSSI
- HC

SUMMARY:
Nonsuicidal self-injury (NSSI) is defined as direct, deliberate bodily harm without suicidal intention. In recent years, growing evidence suggests that NSSI has become a worldwide public health issue. People with NSSI behaviors, especially adolescents, commonly exhibit emotion-related and interpersonal problems. Pain empathy represents an essential basal domain of socio-emotional processing and refers to the ability to empathize, connect and share with others' pain. However, altered empathic processing has not been systematically examined in adolescents with NSSI. To this end, the current functional magnetic resonance imaging (fMRI) study will recruit one group of NSSI adolescents (n=40) and one healthy control (HC) group (n=40), to compare their neural activity regarding pain empathy processing, which is measured by blood oxygenation level-dependent (BOLD) fMRI. The investigators included conditions of physical pain empathy (stimuli depicting noxious stimulation to the limbs) and affective pain empathy (stimuli depicting faces expressing pain) as well as corresponding control stimuli. The investigators hypothesize that compared to HC, NSSI adolescents show increased empathic reactivity to physical pain stimuli in salience and arousal related brain regions but decreased empathic reactivity to affective pain empathic stimuli.

ELIGIBILITY:
Inclusion Criteria:

* 15-18 years
* right-handed
* normal or corrected normal visual acuity
* meet the proposed DSM-5 frequency criteria (e.g., ≥5 days of NSSI behaviors in the past year)

Exclusion Criteria:

* diagnosis of borderline personality disorder, major depressive disorder, other
* psychiatric disorders, etc.
* high suicidal risk
* recent use of medications that can affect neural activity
* have received or are receiving Dialectical Behavior Therapy (DBT) other treatment for emotional problems within the past 6 months
* have a contraindication to MRI scanning (e.g., metal implants, claustrophobia or other conditions that make them inappropriate for MRI scanning)

Ages: 15 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Treatment-seeking NSSI individuals will be recruited from local hospitals and HC from the community
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-12-06 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Neural activity as indexed by BOLD fMRI | About 8 minutes
  Brain activity will be monitored by task-based fMRI. The paradigm will present affective and physical pain empathy pictures and matched control stimuli. Alterations in the patients will be determined by comparing neural activity to the experimental conditions between the experimental groups (NSSI vs. HC) using ANOVA models.

CONTACTS AND LOCATIONS:
Locations (1):
- Sichuan Provincial Center for Mental Health, Sichuan Provincial People's Hospital, University of Electronic Science and Technology of China, Chengdu, Sichuan, China